CLINICAL TRIAL: NCT04663685
Title: MoveStrong at Home: A Feasibility Study of a Model for Remote Delivery of Functional Strength and Balance Training Combined With Nutrition Education for Older Pre-frail Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 42206
Record Dates: First submitted 2020-10-08; First posted 2020-12-11 (Actual); Results first posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2023-11

CONDITIONS: Arthritis; Cancer; Cardiovascular Diseases; Chronic Lung Disease; Congestive Heart Failure; Diabetes; Hypertension; Kidney Diseases; Obesity; Osteoporosis; Stroke; Frailty
Keywords: remote delivery; exercise; pre-frail; nutrition; pilot study
MeSH Terms: conditions — Arthritis; Neoplasms; Cardiovascular Diseases; Heart Failure; Diabetes Mellitus; Hypertension; Kidney Diseases; Obesity; Osteoporosis; Stroke; Frailty; Motor Activity | interventions — Resistance Training; Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: This is an 8-week feasibility study with a 4-week follow-up. Time series design.
  Note: 6-month follow-up was optional and exploratory in nature.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): This was the only arm in the study. All participants were allocated to this arm, where they received an 8-week remotely-delivered exercise and nutrition program.
  Interventions: Other: Exercise program; Other: Nutrition education

INTERVENTIONS:
Other: Exercise program — Participants received two 1-on-1 exercise sessions per week to start. Each session lasted 30 minutes. As progress was made, participants were encouraged to exercise independently outside the structured sessions while continuing to receive a 1-on-1 session each week. The individualized exercises were aligned with functional movements to promote personal relevance: balance, pull, squat, push, hinge, lift & carry and calf raise.
Other: Nutrition education — Participants received a nutrition education booklet and had access to five online videos that correspond to key topics in the booklet (reading nutrition labels, types of protein, foods containing protein, incorporating protein into meals, spreading protein in meals throughout the day). Participants attended three 60-minute nutrition Q&A sessions led by a dietitian, where the group reviewed content from the booklet and videos, and discussed personalized strategies to increase protein intake.

SUMMARY:
Sufficient muscle strength helps to get out of a chair and can prevent falls. Up to 30% of older adults experience age-related loss of muscle strength, which can lead to frailty and health instability. Exercise helps to build muscle, maintain bone density and prevent chronic disease, especially during the aging process. However, more than 75% of Canadian adults ≥18 years of age are not meeting physical activity guidelines. In addition, it is known that malnutrition, including low protein intake, may lead to poor physical function. While there are services to support exercise and nutrition, barriers to implementing them persist. The COVID-19 pandemic has exacerbated the potential for physical inactivity, malnutrition, and loneliness among older adults, especially those with pre-existing health or mobility impairments. Now and in future, alternate ways to promote exercise and proper nutrition to the most vulnerable are needed. The investigators propose to adapt MoveStrong, an 8-week education program combining functional and balance training with strategies to increase protein intake. The program was co-developed with patient advocates, Osteoporosis Canada, the YMCA, Community Support Connections and others. MoveStrong was delivered by telephone or web conference to older adults in their homes, using mailed program instructions, 1-on-1 training sessions through Physitrack®, as well as online nutrition Q&A sessions and group discussion sessions over Microsoft® Teams. The primary aim of this study was to assess feasibility and acceptability of a remote model as determined by recruitment (≥ 25 people in 3 months), retention (≥80%), adherence of (70%) and participant experience.

DETAILED DESCRIPTION:
MoveStrong at Home is an 8-week pilot study with a 4-week follow-up.

The primary research question pertains to the feasibility of implementation, defined by recruitment (number of participants recruited), retention (number retained at follow up), and adherence (percentage of exercise and nutrition sessions completed) and participant experience. The criteria for success included recruitment of 8 participants per month (up to a total of 25 participants in 3 months), retention of ≥80% at follow-up, and adherence of ≥70% across all exercise and nutrition sessions.

For secondary outcomes, the investigators assessed the effects of MoveStrong at Home on physical activity, fatigue, mental health and social isolation, quality of life, as well as protein/energy intake via telephone at baseline, post intervention and at follow-up. The following questionnaires were used: Physical Activity Scale for the Elderly; Centre for Epidemiologic Studies Depression Scale-fatigue questions; Warwick-Edinburgh Mental Well-being Scale; EQ5D5L20; and the Automated Self-Administered 24-Hour Dietary Assessment Tool (via interview). Physical function was assessed at baseline, post intervention and at follow-up using adapted and self-administered versions of the Short Performance Physical Battery balance test and the 30-second chair stand test. Qualitative exit and follow-up interviews were used to capture participant experience and identify barriers and facilitators to implementation and maintenance. The investigators monitored falls and adverse events throughout the study.

The investigators recruited participants in two phases. The investigators recruited 9 participants between October 5th and October 23rd, 2020 to begin the intervention together by November 2020. Participants recruited after that date participated in screening and assessments between November 2020 and January 2021, and began the intervention in January 2021. The investigators considered making modifications to the protocol to address any challenges that arose during delivery with the first phase of participants. Investigators over recruited by 5 participants to account for possible dropouts.

Each participant started the intervention with two 1-on-1 sessions on non-consecutive days (Monday to Friday) and completed the third session on their own. As progress is made, participants continued to receive a 1-on-1 session each week and completed two sessions independently. If a participant was unable to attend a 1-on-1 session due to a prior commitment, illness, or injury, a make-up session was scheduled for the same week or following week as necessary.

In addition, individuals participated in three dietitian-led virtual group Q&A sessions to review content from the booklet and videos, as well as discuss more personalized strategies to increase protein intake. The dietitian considered the cost of preparing high-protein foods and the accessibility of these foods during a time of physical distancing. 60-minute small group seminars (5-10 participants) occurred on weeks 2, 4, and 6 (Wednesday).

An optional group discussion session that focused on behaviour change techniques took place on weeks 3, 5 & 7 (Wednesday). The intention was to foster a sense of community and allow participants to share their experiences with one another. These sessions did not count toward adherence.

The goal of the investigators was not to test the efficacy of exercise, but to evaluate the implementation of a scalable and sustainable models to promote exercise at home or in the community.

ELIGIBILITY:
Inclusion Criteria:

* Has at least one of the following chronic conditions: arthritis, cancer (other than minor skin cancer), cardiovascular disease, chronic lung disease, congestive heart failure, diabetes, hypertension, kidney disease, obesity, osteoporosis, stroke
* Scored ≥ 1 point on the FRAIL Scale
* Able to give informed consent

Exclusion Criteria:

* Current or recent (within the past 6 months)participation in progressive resistance training program ≥ 2 times per week
* Receiving palliative care
* Unable to perform basic activities of daily living or follow 2-step commands (moderate-severe cognitive impairment)
* Upcoming travel plans (travelling> 1 week during the program)
* Absolute exercise contraindications (ACSM guidelines)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lora Giangregorio, PhD, Principal Investigator — University of Waterloo
Locations (1):
- University of Waterloo, Waterloo, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greenwood JL, Joy EA, Stanford JB. The Physical Activity Vital Sign: a primary care tool to guide counseling for obesity. J Phys Act Health. 2010 Sep;7(5):571-6. doi: 10.1123/jpah.7.5.571. PMID 20864751
- [Background] Resnick B, Jenkins LS. Testing the reliability and validity of the Self-Efficacy for Exercise scale. Nurs Res. 2000 May-Jun;49(3):154-9. doi: 10.1097/00006199-200005000-00007. PMID 10882320
- [Background] McAuley E, Mailey EL, Mullen SP, Szabo AN, Wojcicki TR, White SM, Gothe N, Olson EA, Kramer AF. Growth trajectories of exercise self-efficacy in older adults: influence of measures and initial status. Health Psychol. 2011 Jan;30(1):75-83. doi: 10.1037/a0021567. PMID 21038962
- [Background] Bohannon RW. Sit-to-stand test for measuring performance of lower extremity muscles. Percept Mot Skills. 1995 Feb;80(1):163-6. doi: 10.2466/pms.1995.80.1.163. PMID 7624188
- [Background] Jones CJ, Rikli RE, Beam WC. A 30-s chair-stand test as a measure of lower body strength in community-residing older adults. Res Q Exerc Sport. 1999 Jun;70(2):113-9. doi: 10.1080/02701367.1999.10608028. PMID 10380242
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Keller HH, Goy R, Kane SL. Validity and reliability of SCREEN II (Seniors in the community: risk evaluation for eating and nutrition, Version II). Eur J Clin Nutr. 2005 Oct;59(10):1149-57. doi: 10.1038/sj.ejcn.1602225. PMID 16015256
- [Background] Subar AF, Kirkpatrick SI, Mittl B, Zimmerman TP, Thompson FE, Bingley C, Willis G, Islam NG, Baranowski T, McNutt S, Potischman N. The Automated Self-Administered 24-hour dietary recall (ASA24): a resource for researchers, clinicians, and educators from the National Cancer Institute. J Acad Nutr Diet. 2012 Aug;112(8):1134-7. doi: 10.1016/j.jand.2012.04.016. Epub 2012 Jun 15. No abstract available. PMID 22704899
- [Background] Clark RE, Milligan J, Ashe MC, Faulkner G, Canfield C, Funnell L, Brien S, Butt DA, Mehan U, Samson K, Papaioannou A, Giangregorio L. A patient-oriented approach to the development of a primary care physical activity screen for embedding into electronic medical records. Appl Physiol Nutr Metab. 2021 Jun;46(6):589-596. doi: 10.1139/apnm-2020-0356. Epub 2020 Nov 23. PMID 33226847
- [Background] Radloff, LS. The CES-D scale: A self-report depression scale for research in the general population. Applied psychological measurement,1977; 1(3), 385-401.
- [Background] Xie F, Pullenayegum E, Gaebel K, Bansback N, Bryan S, Ohinmaa A, Poissant L, Johnson JA; Canadian EQ-5D-5L Valuation Study Group. A Time Trade-off-derived Value Set of the EQ-5D-5L for Canada. Med Care. 2016 Jan;54(1):98-105. doi: 10.1097/MLR.0000000000000447. PMID 26492214
- [Result] Wang E, Keller H, Mourtzakis M, Rodrigues IB, Steinke A, Ashe MC, Thabane L, Brien S, Funnell L, Cheung AM, Milligan J, Papaioannou A, Weston ZJ, Straus S, Giangregorio L. MoveStrong at home: a feasibility study of a model for remote delivery of functional strength and balance training combined with nutrition education for older pre-frail and frail adults. Appl Physiol Nutr Metab. 2022 Dec 1;47(12):1172-1186. doi: 10.1139/apnm-2022-0195. Epub 2022 Sep 15. PMID 36108334

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were primarily recruited from email or telephone contact lists. In addition, we asked colleagues and collaborators to forward the link to potential participants on their distribution lists. Research support staff and Kinesiologists at two Schlegel Villages and one Luther Villages recruited participants using flyers and word of mouth. The recruitment period went from October 5th, 2020, to December 28th, 2020.
Period: Overall Study
Arm/Group | Single Arm
Started | 30
Completed | 28
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Modified PROGRESS-Plus Framework.
Arm/Group | Single Arm
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] — Average Age and Standard Deviation
  years | 74 (7)
Sex/Gender, Customized [Number; unit: participants] — Biological Sex
  participants
    Female | 26
    Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Self-identified ethnicity
  Participants
    Caucasian | 29
    South Asian | 1
Region of Enrollment [Count of Participants; unit: Participants] — Recruitment was restricted to Ontario, Canada residents.
  Participants
    Canada | 30

OUTCOME MEASURES:

1. Primary Outcome: Recruitment
Description: The number of participants recruited >25.
Time Frame: Through study completion, an average of 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 30
Participants | 30

2. Primary Outcome: Retention
Description: Feasibility threshold: The number of participants retained at follow-up >80%.
Time Frame: Through study completion, an average of 12 weeks
Population: 2 participants withdrew from the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 30
Participants | 28

3. Primary Outcome: Average Adherence to Nutrition Sessions
Description: Participants were encouraged to attend 3 nutrition sessions that took place on weeks 2, 4 and 6 of the intervention (12 weeks).
  Feasibility threshold: "Attendance" or the average proportion of nutrition sessions >67% or >2/3 sessions.
Time Frame: Through study completion, an average of 12 weeks
Population: 2 participants withdrew from the intervention.
Measure: Mean (Standard Deviation); unit: sessions
Units Other Than Participants: sessions
Arm/Group | Single Arm
Number analyzed (Participants) | 28
Number analyzed (sessions) | 3
sessions | 2.5 (0.5)

4. Primary Outcome: Average Adherence to Exercise Sessions
Description: Participants were encouraged to complete at least 3 exercise sessions per week (one supervised and two independent) for the duration of the intervention (12 weeks).
  Feasibility threshold: "Attendance" or the average proportion of exercise sessions completed >70% or 25.3/36 sessions.
Time Frame: Through study completion, an average of 12 weeks
Population: 2 participants withdrew from the intervention.
Measure: Mean (Standard Deviation); unit: sessions
Units Other Than Participants: number of sessions
Arm/Group | Single Arm
Number analyzed (Participants) | 28
Number analyzed (number of sessions) | 36
sessions | 30.2 (6.5)

5. Secondary Outcome: Physical Activity
Description: A Physical Activity Screen (PAS) was used to capture average minutes of moderate-to-vigorous physical activity each week (Clark et al., 2020). This tool was created based on questions used by Exercise is Medicine in the Physical Activity Vital Sign questionnaire (Greenwood et al., 2010). The results were compared to national exercise guidelines for older adults that promote ≥150 minutes and ≥2 session of muscle strengthening per week. A higher score indicated a better outcome.
Time Frame: Baseline, week 9, week 12
Population: 2 participants withdrew from the intervention.
Measure: Mean (Standard Deviation); unit: weekly minutes of physical activity
Arm/Group | Single Arm
Number analyzed (Participants) | 28
weekly minutes of physical activity
  Baseline | 180 (82)
  End of the study: number analyzed (Participants) | 27
  End of the study | 310 (85)
  Follow-up: number analyzed (Participants) | 27
  Follow-up | 263 (71)

6. Secondary Outcome: Exercise Self-efficacy Scale
Description: A modified version of the Exercise Self-Efficacy Scale (ESES) was used to assess levels of planning and execution of exercise related activities (Resnick & Jenkins, 2000). There were a total of 11 questions. The lowest response option to each question was "Not true at all = 1", while the highest was "Exactly true = 5". Responses closer to the highest response option indicate a better outcome. Overall instrument score ranged from 11-55 points.
Time Frame: Baseline, week 9, week 12
Population: 2 participants withdrew from the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale of 11-55
Arm/Group | Single Arm
Number analyzed (Participants) | 28
score on a scale of 11-55
  Baseline | 26.4 (5.2)
  End of the study | 33.6 (5.3)
  Follow-up | 35.0 (5.6)

7. Secondary Outcome: 30-second Chair Stand
Description: The 30-second Chair Stand was used to access lower extremity muscle function (Bohannon, 1995; Jones et al., 1999). The instructions for this test were adapted for self-administration under the remote supervisor supervision of the exercise physiologist. A higher score on the test indicated a better outcome.
Time Frame: Baseline, week 9, week 12
Population: 2 participants withdrew from the intervention.
Measure: Mean (Standard Deviation); unit: number of chair stands completed in 30s
Arm/Group | Single Arm
Number analyzed (Participants) | 28
number of chair stands completed in 30s
  Baseline | 8.00 (2.41)
  End of study | 11.50 (2.72)
  Follow-up | 12.54 (2.81)

8. Secondary Outcome: Static Balance
Description: Static balance was measured using Short Performance Physical Battery (SPPB) (J. M. Guralnik et al., 1994) balance subscale. The subscale scores ranged from 0-4, with a higher score indicating greater balance. The instructions for this test were adapted for self-administration under the remote supervisor supervision of the exercise physiologist.
  Please note that the SPPB gait speed and chair stand subscales were not included as a part of the assessment. Therefore the total score for the SPPB (0-12) was not summed.
Time Frame: Baseline, week 9, week 12
Population: 2 participants withdrew from the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 28
score on a scale
  Baseline | 3.54 (0.39)
  End of study | 3.64 (0.39)
  Follow-up | 3.82 (0.26)

9. Secondary Outcome: Fatigue
Description: Fatigue was assessed using the Center for Epidemiologic Studies Depression Scale-fatigue questions (CES-D) (Radloff, 1977). Only two questions on the CES-D were used: "I felt that everything I did was an effort" and "I could not get going". Scores ranged from of 0-6 and were summed from the two selected questions (lowest response option was "Rarely (<1 day) = 0", highest response option was "Nearly every day = 3"). Responses closer to the lowest response option indicated a better outcome.
Time Frame: Baseline, week 9, week 12
Population: 2 participants withdrew from the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 28
score on a scale
  Baseline | 1.86 (0.53)
  End of study | 1.07 (0.41)
  Follow-up | 1.14 (0.46)

10. Secondary Outcome: Mental Health and Social Isolation
Description: The Warwick-Edinburgh Mental Well-being Scale (WEMWBS) was used to assess positive aspects of mental health. Score ranges from 14-70 and were summed from 14 questions (lowest response option was "None of the time =1", highest response option was "All of the time = 5"). Responses closer to the highest response option indicated a better outcome.
Time Frame: Baseline, week 9, week 12
Population: 2 participants withdrew from the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 28
score on a scale
  Baseline | 53.5 (3.4)
  End of study | 54.8 (3.0)
  Follow-up | 53.5 (3.5)

11. Secondary Outcome: Quality of Life Score
Description: The EuroQol Group 5 Dimension 5 Level (EQ5D5L) questionnaire was used to evaluate health-related quality of life (Herdman et al., 2011). The system comprised five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension had five levels: "no problems = 1" to "extreme problems = 5". Responses with lower scores indicated a better outcome. An index value ranging from 0-1 is then generated from the equation by from the scores of the five domains (Xie et al. 2016)
Time Frame: Baseline, week 9, week 12
Population: 2 participants withdrew from the intervention.
Measure: Mean (Standard Deviation); unit: index value/scores on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 28
index value/scores on a scale
  Baseline | 0.832 (0.024)
  End of study | 0.805 (0.034)
  Follow-up | 0.807 (0.038)

12. Secondary Outcome: Nutritional Risk
Description: The SCREEN tool is a valid and reliable nutrition questionnaire designed specifically for older adults (Keller et al., 2005). This tool was used to assess appetite, understand eating habits, and record recent changes in weight. Scores ranged from of 0-64 and were summed from 14 questions (lowest response option was "0", highest response option was "4"). Responses closer to the highest response option indicated a better outcome.
Time Frame: Baseline, week 9, week 12
Population: 2 participants withdrew from the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 28
score on a scale
  Baseline | 30.9 (2.5)
  End of study | 40.3 (2.7)
  Follow-up | 38.8 (3.3)

13. Secondary Outcome: Dietary Protein Intake
Description: ASA24®-Canada was a guided web-based tool used to record a three 24-hour diet recalls. All food and drinks consumed by the participant on two weekdays and one weekend day (3 days in total) were reported to track protein intake (Subar et al., 2012). An average of the three days was then calculated.
Time Frame: Baseline, week 9, week 12
Population: 2 participants withdrew from the intervention.
Measure: Mean (Standard Deviation); unit: grams of dietary protein
Arm/Group | Single Arm
Number analyzed (Participants) | 28
grams of dietary protein
  Baseline | 79.8 (9.6)
  End of study | 92.7 (11.7)
  Follow-up | 89.0 (11.5)

ADVERSE EVENTS:
Time Frame: From baseline to 12 weeks of the intervention
Description: Health Canada Definition
  Public Health Agency of Canada (2018) Reporting Adverse Reactions to Marketed Health Products - Guidance Document for Industry, Ministry of Health. Available at: https://www.canada.ca/en/health-canada/services/drugs-health-products/reports-publications/medeffect-canada/reporting-adverse-reactions-marketed-health-products-guidance-industry.html
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 5/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=28)
Non-serious, non-attributed (Musculoskeletal and connective tissue disorders) | 5 (6) — Participants were asked on a weekly basis (at the start of 1-on-1 exercise sessions). We reported all serious and non-serious adverse events and identified those attributed to intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT04663685/Prot_SAP_ICF_000.pdf